CLINICAL TRIAL: NCT03447210
Title: Integrating Assisted Partner Services and Phylogenetics for HIV and HCV Prevention
Brief Title: Study of HIV, HCV, APS and Phylogenetics for PWID
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Kenyatta National Hospital (Other Government); Kenya Ministry of Health (Other Government); University of KwaZulu (Other)
Responsible Party: Principal Investigator, Carey Farquhar, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001536; R01DA043409 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: HIV/AIDS; Hepatitis C
Keywords: Persons who inject drugs (PWID); Phylogenetics; HIV testing; HCV testing; HIV care cascade; Assisted partner services
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Prospective cohort study with nested cross-sectional studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assisted Partner Services (Experimental): All participants in this arm will be offered assisted partner services (APS) which involves outreach to sexual partners and to individuals with whom they use injection drugs. When partners are contacted they are offered HIV and HCV testing. There is no comparison arm.
  Interventions: Behavioral: Assisted Partner Services

INTERVENTIONS:
Behavioral: Assisted Partner Services — Contact tracing for sexual and drug-sharing partners to notify about exposure to HIV and offer HIV and hepatitis C testing with linkage to care and partner services for those who test positive.

SUMMARY:
This study will determine whether assisted partner notification services (APS) can identify and link to care, the sexual and needle-sharing partners of HIV-infected and HIV/hepatitis C (HCV) co-infected persons who inject drugs (PWID). It will also define the risk factors for onward HIV and HCV transmission among PWID using viral phylogenetics.

DETAILED DESCRIPTION:
Overview: This NIH-funded study uses assisted partner services (APS) to identify HIV-infected and HCV-infected persons who inject drugs (PWID) in Kenya and link them to care. In addition to determining the role of APS in HIV and HCV case-finding for this hard-to-reach key population, we leverage our experience with HIV and HCV phylogenetics in the US and South Africa to define modes and risk factors for onward viral transmission. The specific aims of the proposal are as follows:

AIM 1. To determine whether contact tracing and partner notification practices, known in Kenya as assisted partner services (APS), can identify and link to care, the sexual and injection partners of HIV-infected and HIV/ hepatitis C (HCV) co-infected persons who inject drugs (PWID).

AIM 2. To define the risk factors for HIV transmission among PWID, and to elucidate the role of PWID in the overall Kenyan HIV epidemic, using viral genetic sequencing techniques.

AIM 3. To characterize the modes and risk factors for onward HCV transmission among PWID using viral genetic sequencing.

Design: We will enroll 1000 HIV-infected PWID through a needle and syringe exchange program (NSP) in Nairobi, Kenya. Each index participant will undergo a structured questionnaire, a rapid HCV test, a blood draw, and will provide locator information regarding their sexual and injection partners from the past 3 years. Study staff will then attempt to locate all partners. Once located, partner participants will undergo rapid HIV and HCV testing, a structured questionnaire, and a blood draw. All blood samples will be sent to a central laboratory in Nairobi for processing. Dried blood spot samples will be created in Nairobi and will later be sent to the University of KwaZulu-Natal for quantitative viral loads for both HIV and hepatitis C, and follow-up phylogenetic testing. All participants who test positive for HIV or hepatitis C will be referred for counseling and treatment. HIV care and treatment will take place at multiple local centers offering these services.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age
* Active intravenous drug use (IDU) as defined by injecting at least twice in the past month
* Willing and able to provide informed consent
* HIV infected (either new diagnosis or known diagnosis)
* Willing and able to provide locator information for sexual and/or injecting partners

Exclusion Criteria:

• Classified as at high risk for IPV*

*Participants will be classified as at moderate risk for IPV if they report 1) history of IPV during their lifetime either from a current or past partner; and/or 2) fear of IPV if they participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4301 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Sexual partners tested | 4 years
  Numbers of sexual partners tested for HIV and HCV per index participant
Injecting partners tested | 4 years
  Numbers of injecting partners tested for HIV and HCV per index participant
Partners diagnosed with HIV and HCV | 4 years
  Number of partners newly diagnosed with HIV and HCV infection per index case
HIV-infected partners linked to HIV care | 4 years
  Percentage of HIV-infected partners linked to HIV care
HCV-infected partners linked to HCV care | 4 years
  Percentage of HCV-infected partners linked to HCV care
Index participants linked to HIV and HCV care | 4 years
  Percentage of index participants linked to HIV and HCV care

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Herbeck, PhD, Principal Investigator — University of Washington; Carey Farquhar, MD, MPH, Principal Investigator — University of Washington
Locations (3):
- Kenya (3):
  - Githurai Drop-in Centre, Nairobi
  - Ngara Health Centre, Nairobi
  - Pangani Drop-in Centre, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
The proposed studies will include the following data: self-reported demographic and behavioral data, medical/sexual histories, HIV/HCV test results, and HIV/HCV genetic sequences. To facilitate the data sharing process, we will consider the need for data sharing in the study design, creation of informed consent documents, and the structure of data collection. Release of completed viral gene sequences (on NCBI Genbank) shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5-10 years

REFERENCES:
- [Derived] Monroe-Wise A, Mbogo L, Guthrie B, Bukusi D, Sambai B, Chohan B, Scott J, Cherutich P, Musyoki H, Bosire R, Dunbar M, Macharia P, Masyuko S, Wilkinson E, De Oliveira T, Ludwig-Barron N, Sinkele B, Herbeck J, Farquhar C. Peer-mediated HIV assisted partner services to identify and link to care HIV-positive and HCV-positive people who inject drugs: a cohort study protocol. BMJ Open. 2021 Apr 24;11(4):e041083. doi: 10.1136/bmjopen-2020-041083. PMID 33895711